CLINICAL TRIAL: NCT05473949
Title: Ketofol (Ketamine and Propofol) Versus Propofol for Sedation in Cholangiopancreatography for ASA III and ASA IV Patients
Brief Title: Ketofol Versus Propofol for Sedation in Cholangiopancreatography for ASA III and ASA IV Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar Universitário Lisboa Norte (Other)
Responsible Party: Principal Investigator, Henrique Xavier Ornelas Gouveia, Principal Investigator, Centro Hospitalar Universitário Lisboa Norte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 566/15
Record Dates: First submitted 2022-03-28; First posted 2022-07-26 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): ASA Standard monitorization and nasal spectacle capnography (OC) were used. Supplementary supply of O2 is placed at 2-3 L/min also by OC.
  The drugs were randomized of the study begins. The investigators didn't know whether ketamine is present in syringes prepared with propofol or not, acting in the same way for both drug combinations.
  Sedation was performed with:
  1. Propofol: induction with a bolus of 1% propofol (10mL syringe) administered at a dose of 0.75mg/kg; maintenance with 1% propofol infusion (20mL syringe), at an infusion rate of 6-7mg/kg/h.
  In both arms:
  * 4 mg of I.V. dexamethasone were administered.
  * At the beginning of the procedure and atropine and ephedrine were prepared.
  * At the end of the procedure, paracetamol I.V. 15mg/kg was administered.
  * If the patient reports VAS>3 pain in recovery, metamizole magnesium 15mg/kg is also administered.
  * In case of post-procedure nausea and/or vomiting, 4 mg of ondansetron would be administered as a rescue.
  Interventions: Drug: Profofol for Sedation in Cholangiopancreatography for ASA III and ASA IV Patients
- Ketofol (Active Comparator): 2. Sedation with ketofol in a 1:4 dilution: induction of sedation with bolus of ketofol (dilution containing 9.5 mL of 1% propofol + 0.5 mL of 5% ketamine) (10mL syringe), administered at a dose of 0.75 mg/kg; maintenance with ketofol infusion (dilution containing 19 mL of 1% Propofol + 1 mL of 5% Ketamine), (20mL syringe), at an infusion rate of 6-7mg/kg/h.
  The dose used for bolus induction of sedation in both arms of the study is titrated to the needs of each individual patient, although the target approximates the usual recommended dose. If a propofol or ketofol syringe is insufficient considering the patient's weight, another syringe will be prepared with exactly the same dilution as the first.
  The study was always blind to the investigators.
  Interventions: Drug: Ketofol for Sedation in Cholangiopancreatography for ASA III and ASA IV Patients

INTERVENTIONS:
Drug: Profofol for Sedation in Cholangiopancreatography for ASA III and ASA IV Patients — Use of 1% Propofol (Indution dose: 0.75mg/kg Maintenance dose: 6-7mg/kg/h) for Sedation in Cholangiopancreatography for ASA III and ASA IV Patients
  Arms: Propofol
Drug: Ketofol for Sedation in Cholangiopancreatography for ASA III and ASA IV Patients — use of Ketofol (1% Propofol + 5% Ketamine with a ratio 1/4) Indution dose: 0.75mg/kg Maintenance dose: 6-7mg/kg/h) for Sedation in Cholangiopancreatography for ASA III and ASA IV Patients
  Arms: Ketofol

SUMMARY:
This study is a double blind randomized controlled trial. The investigators randomized ASA III and IV patients who underwent cholangiopancreatography. The investigators gave Propofol or Ketofol and compared the outcomes. The primary outcome was security (respiratory depression / hypoventilation).

DETAILED DESCRIPTION:
Randomization is performed by the nurse responsible for preparing the anesthesia drugs. The nurse randomly removes an envelope from a previously prepared container with as many envelopes as the number of patients calculated for the sample. Each envelope, which will be sealed, contains the branch to which the patient belongs (propofol or ketofol) and instructions for the preparation of the respective drugs.

The sample was calculated for a significance level of 5% and a test power of 95%, assuming that, on average, the primary outcome of this study - respiratory depression - is observed in 3% of the population undergoing sedation with ketofol and to 25% of patients undergoing sedation with propofol. The result of the calculation includes 51 patients for each branch of the study (considering the one-tailed hypothesis test).

Data collection is expected to take place over 5 months, taking place between October 2016 and March 2017.

The study is designed to be blinded to the patient and the anesthesiologist/investigator.

The anesthesia nurse, after preparing the drugs according to the instructions on the envelope containing the branch of the study to which the patient belongs, should label each syringe in a non-committal manner.

Statistical analysis was performed using the IBM SPSS Statistics 27.

It will not be necessary to resort to the monitoring committee, since no method or technique different from the one usually practiced will be applied

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* ASA III and IV
* Submitted to retrograde cholangiopancreatography

Exclusion Criteria:

* Patient refuse
* ASA I, II and V
* Ketamine contraindications
* Allergies to Propofol, Ketamine, dexamethasone, paracetamol, metamizole, ondanseteon or other.
* General anesthesia necessary I
* Incapacitaty to sign or absence of patient legal representation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Security - Hypoventilation / Respiratory Depression | Intraprocedure
  Hypoventilation / Respiratory Depression defined as: Need for airway management (mandibular subluxation or other permeabilization maneuvers, use of adjuvants, need for assisted or controlled ventilation); Oxygen desaturation measured by pulse oximeter n(<95%); Apnea (>10 seconds)

SECONDARY OUTCOMES:
Security - Intraprocedure hypotension | During the procedure and immediately after the end of procedure
  Intraprocedure hypotension defined as: non invasive arterial systolic pressure < 90 mmHg and/or diastolic < 60 mmHg OR non invasive arterial pressure < 20% of the base value
Efficiency - Intraprocedure opioid necessity | During the procedure and immediately after the end of procedure
  Intraprocedure opioid necessity: Pain during the procedure, interpreted by the anesthesiologist through patient complaints or through analysis of hemodynamic parameters; Pain after the procedure, quantified by the visual analogue pain scale (VAS) 0-10, where 0 corresponds to no pain and 10 corresponds to the worst possible pain); Need for supplemental analgesia.
Efficiency - Assessment of sedation level | During the procedure and immediately after the end of procedure
  Assessment of sedation level : the investigators measured the level of sedation for each participant with the Sedation Ramsay Scale.
Quality - Patients satisfaction | At the end of the procedure (when the patient lucid and oriented in person, time and space) and 24 hours after the end of the procedure
  Patients satisfaction at the end of the procedure and after 24 hour: the investigators evalueted the patient satisfaction with a 4 point rating scale (1 - dissatisfied, 2- little satisfied, 3- satisfied, 4- very satisfied); and no opinion (NP). This evalution was perfomed after gaining consciousness (being oriented in the person, time and space) in the first two hours after the end of the procedure.
  The patient was contacted 24 hours after the end of the procedure (by phone or in person if still hospitalized) by one of the investigators, in order to assess the patient's well-being, degree of pain, occurrence of nausea or vomiting and satisfaction at the time. These data are recorded in a specific form, which again does not specify which branch of the study the patient was assigned to (blind to the investigator), and stored in a separate folder with the same numerical code assigned to the form completed the day before by the investigators.
Quality - Gastroenterologist satisfaction | Immediately at the end of the procedure
  Gastroenterologist satisfaction: the investigators evalueted the Gastroenterologist satisfaction at the end of the procedure with a 4 point rating scale (1 - dissatisfied, 2- little satisfied, 3- satisfied, 4- very satisfied); and no opinion (NP).
Quality - Occurrence of postoperative nausea or vomiting | In the first 24 hours after the end of the procedure
  Occurrence of postoperative nausea or vomiting: the investigators recorded the occurrence of nausea or vomiting after the procedure within the first 24 hours.
Quality - Occurence of psychotomimetic effects | In the first 24 hours after the end of the procedure
  Occurence of psychotomimetic effects: the investigators recorded the occurrence of psychotomimetic effects after the procedure within the first 24 hours.
  The investigators verify the occurrence of the most frequent psychomimetic symptoms by questionnaire and medical/physical evaluation (anxiety, confusion, disorientation / psychomotor agitation, dysphoria, dissociative state and delirium with or without hallucinations, abnormal dreams, nightmares, insomnia)

CONTACTS AND LOCATIONS:
Overall Officials: Amélia Almeida, Study Chair — Centro Hospitalar e Universitário de Lisboa Norte

IPD SHARING:
Plan to Share IPD: No
Approval from other investigators is required and research center approval - Centro Hospitalar e Universitário de Lisboa Norte

REFERENCES:
- [Background] Standard for basis anesthetic monitoring - Committee of Origin: Standards and Practice Parameters; Approved by the ASA House of Delegates on October 21, 1986, and last amended on October 20, 2010 with an effective date of July 1, 2011
- [Background] Statement on nonoperating room anesthetizing locations - Committee of origin: Standards and Practice Parameters; Approved by the ASA House of Delegates in October 19,1994, and last amended on October 16, 2013
- [Result] Green SM, Andolfatto G, Krauss B. Ketofol for procedural sedation? Pro and con. Ann Emerg Med. 2011 May;57(5):444-8. doi: 10.1016/j.annemergmed.2010.12.009. Epub 2011 Jan 14. No abstract available. PMID 21237532
- [Result] Ronald D. Miller, Miller's Anesthesia, 7th edition, Section III - Anesthetic Pharmacology, Chapter 26: Intravenous Anesthetics, p. 724